CLINICAL TRIAL: NCT04461080
Title: Screening for Poverty And Related Social Determinants and Intervening to Improve Knowledge of and Links to Resources (SPARK): a Randomized Controlled Study
Brief Title: Screening for Poverty And Related Social Determinants to Improve Knowledge of and Links to Resources (SPARK)
Acronym: SPARK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Memorial University of Newfoundland (Other); Dalhousie University (Other); University of Manitoba (Other); University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UpstreamLab2020-1
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Poverty
Keywords: poverty; income; social determinants of health
MeSH Terms: interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: parallel, two-arm 1:1 individual participant allocation randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated care promoter (Experimental): Patients who are randomized to the intervention group will be connected with a trained Community Health Worker (CHW). The CHW is a peer with lived-experience of system navigation that could have a background in social work, health promotion or community work. All CHWs will receive 2 weeks of training to assist participants with social needs.
  Interventions: Behavioral: Community Health Worker
- Information on community resources (Active Comparator): Patients randomized to the control group will receive a list of tailored written information.
  Interventions: Behavioral: Community Health Worker

INTERVENTIONS:
Behavioral: Community Health Worker — Trained Community Health Worker

SUMMARY:
The SPARK RCT will test the impact of engagement with a Community Health Worker who is embedded in interprofessional primary care teams on change in estimated annual income at 6 months for people living in poverty.

DETAILED DESCRIPTION:
Population: Patients seen by interprofessional primary care teams who are living on estimated annual incomes that are below the Canadian Low-Income Cut-Off (LICO)

Intervention: A Community Health Worker who implements an intervention that addresses a number of social needs, including improving income security, access to prescription medications, access to housing, reducing social isolation, paying for utilities and access to transportation

Control: Information on community resources on social needs

Outcome: Change in estimated annual income between baseline and at 6 months

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old AND live in a household with an income below the Low-Income Cut-OFF AND agree to receive assistance with social needs

Exclusion Criteria:

* Has worked with a similar CHW or intervention in the past 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We will ask participants both their sex assigned at birth and their current gender identity, and offer a number of options.
Enrollment: 110 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
change in estimated annual income | 6 months
  The primary outcome will be change in estimated annual income, assessed at baseline and at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Pinto, MD MSc, Principal Investigator — University of Toronto

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be made available to qualified researchers with academic interest in primary care health equity research. Data will only be made available to interested parties after all applicable agreements have been executed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Requests to access the data can be made beginning 3 months and up until 2 years after article publication.
Access Criteria: Access to study IPD will be granted to qualified researchers upon approval of their Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). To submit a request or for any additional questions, please contact Upstreamlab@unityhealth.to.
URL: https://upstreamlab.org/project/spark/

REFERENCES:
- See also: Website for the SPARK Study — https://upstreamlab.org/project/spark/